CLINICAL TRIAL: NCT04151355
Title: The Effect of Atorvastatin on The Prevention of 5-fluorouracil-induced Mucositis in Colorectal Cancer Patients
Brief Title: Effect of Atorvastatin on 5-Fluorouracil Induced Mucositis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Collaborators: Nasser Institute For Research and Treatment (Other Government)
Responsible Party: Principal Investigator, Radwa Salah Lotfy Abdel-Rahman, Clinical Pharmacist at nasser institute, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 216
Record Dates: First submitted 2019-10-28; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, controlled, open-label pilot study will be conducted on 100 colon cancer patients receiving 5-FU adjuvant FOLFOX -6 & FOLFIRI-6 therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin group (Experimental): 50 colorectal cancer patients receiving FOLFOX 6: (Oxaliplatin 85mg/m2 IV over 2 hrs + leucovorin 400mg/m2 IV over 2 hrs, followed by 5-FU 400mg/m2 IV bolus, followed by 5-FU 1,200mg/m2 /day IV x 2 days (total 2,400mg/m2 ) as a 46-48 hr continuous infusion. Repeat every 2 weeks) in addittion to atorvastatin (20 mg once daily) or FOLFIRI 6:( Irinotecan 180mg/m2 IV + leucovorin 400mg/m2 IV, followed by 5-FU 400mg/m2 IV bolus, followed by 5-FU 1,200mg/m2 /day IV x 2 days (total 2,400mg/m2 ) as a 46-48 hr continuous infusion. Repeat every 2 weeks) in addittion to atorvastatin (20 mg once daily) in addittion to atorvastatin (20 mg once daily)
  Interventions: Drug: Atorvastatin 20mg
- Control group (No Intervention): 50 colorectal cancer patients receiving FOLFOX 6: (Oxaliplatin 85mg/m2 IV over 2 hrs + leucovorin 400mg/m2 IV over 2 hrs, followed by 5-FU 400mg/m2 IV bolus, followed by 5-FU 1,200mg/m2 /day IV x 2 days (total 2,400mg/m2 ) as a 46-48 hr continuous infusion. Repeat every 2 weeks) or FOLFIRI 6:( Irinotecan 180mg/m2 IV + leucovorin 400mg/m2 IV, followed by 5-FU 400mg/m2 IV bolus, followed by 5-FU 1,200mg/m2 /day IV x 2 days (total 2,400mg/m2 ) as a 46-48 hr continuous infusion. Repeat every 2 weeks)

INTERVENTIONS:
Drug: Atorvastatin 20mg — atorvastatin (20 mg once daily)
  Arms: Atorvastatin group

SUMMARY:
5-Fuorouracil (5-Fu) remains one of the most effective and most commonly used drugs to treat colorectal cancer. Mucositis is a major complication that occurs in approximately 80% of patients receiving 5-FU and results in abdominal bloating as well as vomiting and diarrhea. oral mucositis (OM) are often very painful and compromise nutrition and oral hygiene as well as increase risk for local and systemic infection.

OM is characterized by an intense inflammatory reaction on the mucosa lamina propria cells, which results in activation of the transcription factor NF-kB. The activation of NF-kB leads to transcription of genes involved in the synthesis of pro-inflammatory cytokines, such as IL-1β, IL-6 and TNF-α. Agents known to attenuate the expression of cytokines have demonstrated efficacy in the prevention of experimental mucositis.

The use of atorvastatin were associated with reduced production of TNF-α and IL-1β and decreased neutrophil infiltration evidenced by histopathological analysis and Myeloperoxidase (MPO) activity. In addition, atorvastatin also reduced oxidative stress and induced an increase in non-protein sulfhydryl groups showing anti-inflammatory and immunomodulatory action.

DETAILED DESCRIPTION:
Chemotherapy has life-threatening or distressing side effects such febrile neutropenia, infections, mucositis, nausea, vomiting, fatigue. Mucositis is deﬁned as inﬂammatory and/or ulcerative lesions of the oral and/or gastrointestinal tract that can be caused by high dose chemotherapy, Infectious disease, immune deﬁciency and medications..

Lesions of oral mucositis (OM) are often very painful and compromise nutrition and oral hygiene as well as increase risk for local and systemic infection. Mucositis can also involve other areas of the alimentary tract; for example, gastrointestinal (GI) mucositis can manifest as diarrhea. Thus, mucositis is a highly significant and sometimes dose-limiting complication of cancer therapy.

OM leads to an increased risk of microbial infections and often entails parenteral nutrition, long-lasting intake of analgesics and extended hospitalization periods. This causes substantial costs to the health system and, also has a considerable impact on the patient's quality of life. Furthermore, dose reduction might become necessary, which limits the efficacy of the antitumor therapy.

OM is characterized by an intense inflammatory reaction on the mucosa lamina propria cells, which results in activation of the transcription factor NF-kB. The activation of NF-kB leads to transcription of genes involved in the synthesis of pro-inflammatory cytokines, such as IL-1β, IL-6 and TNF-α, and agents known to attenuate the expression of cytokines have demonstrated efficacy in the prevention of experimental mucositis.

Conventional chemotherapeutic drugs most frequently associated with mucositis include antimetabolites, such as 5-fluorouracil (5-FU), methotrexate, and purine antagonists. Anthracycline antitumor antibiotics (eg, doxorubicin) and taxanes (eg, paclitaxel and docetaxel) are other chemotherapeutic drugs that commonly cause mucositis.

Over the last five decades, 5-fluorouracil (5-Fu) remains one of the most effective and most commonly used drugs to treat colorectal cancer. The commonly side effects of 5-FU include myelosuppression, dermatitis, cardiac toxicity, diarrhea, and mucositis. Among these adverse effects, gastrointestinal mucositis is a major complication that occurs in approximately 80% of patients receiving 5-FU and results in abdominal bloating as well as vomiting and diarrhea. 5-FU induces inflammation in the small intestine, characterized by the increased intestinal wall thickness and crypt length, the decreased villus height, and the increased myeloperoxidase (MPO) activity in tissues and pro-inflammatory cytokine production in sera..

Statins are potent inhibitors of cholesterol biosynthesis and have been shown to decrease mortality from cardiovascular disease. In addition to their lipid lowering properties by inhibiting 3-hydroxy-3-methylgluteryl coenzyme A (HMG CoA) reductase. Statins possess various pleiotropic effects that include improvement in endothelial dysfunction, increased expression of endothelial nitric oxide synthase (eNOS), enhanced bioavailability of nitric oxide (NO), potent antioxidant potential and anti-inflammatory properties.

It has been reported that simvastatin had significant preventive effects on esophageal, gastric and intestinal damage in a rat model using 10 mg / Kg of simvastatin microemulsion by gavage, beginning one week prior to treatment with MTX, and during treatment with this drug. Animals received i.p. injection of atorvastatin (ATV; 1 or 5 mg/kg), saline or saline/ethanol 30 min before 5-FU and daily for 5 days (5 days) or 10 days (10 days). in hamsters showing significant reduction the macroscopic and micro-scopic lesions induced by 5-FU in the OM of hamsters.

The macroscopic protective effects of atorvastatin were associated with reduced production of TNF-α and IL-1β and decreased neutrophil infiltration evidenced by histopathological analysis and Myeloperoxidase (MPO) activity. In addition, atorvastatin also reduced oxidative stress and induced an increase in non-protein sulfhydryl groups showing anti-inflammatory and immunomodulatory action.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>18 years old).
2. Colon cancer patients ???? who will receive adjuvant FOLFOX 6& FOLFIRI 6 for 6 cycles.
3. ECOG performance status 0-2
4. Adequate bone marrow function (white blood count ≥4,000/mm3, platelet count ≥100,000/mm3), liver function (serum total bilirubin <1.5 mg/dl), renal function (creatinine <1.5 mg/dl).

Exclusion Criteria:

1. Patients who have Clinical GIT mucositis or Periodontal disease.
2. Patients with other primary malignancy.
3. Patients receiving mTOR inhibitors (eg, rapamycin, everolimus, and temsirolimus), EGFR inhibitors (eg, bevacizumab and erlotinib) and tyrosine-kinase inhibitors (eg, sorafenib and sunitinib).
4. Hypersensitivity to Atorvastatin.

6-Pregnant and lactating women. 7- Patients treated with ATV for any other indication. 8- Patient who already have a mucositis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
incidence of mucositis | 6 months
  screening the patients seeking mucositis & grading mucositis using Common Terminology Criteria for Adverse Events, CTCAE version 5 ( ranging from grade 1 of better outcome to 5 of worst outcome ) and evaluating the effect of atorvastatin on mucositis

SECONDARY OUTCOMES:
grade of mucositis | 6 month
  the grade of mucositis will be assessed using common terminology criteria of adverse effects version 5
Pain score | 6 month
  the pain due to mucositis will be assessed using visual analogue scale
Effect of mucositis on patient's daily life | 6-months
  The Oral Health Impact Proﬁle-14 (OHIP-14) will be used to assess the effect of mucositis on the patients' liferanging from 0 of better outcome to 56 of worst outcome
liver function test | 6 months
  serum ALT and AST will be assessed before each cycle
serum levels of tumor necrosis factor α (TNF-α) | 6 months
  serum tumor necrosis factor α (TNF-α) will be assessed at baseline and after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Radwa S. Gad, diplome, Principal Investigator — clinical pharmacist
Locations (1):
- Faculty of Pharmacy, Cairo, Egypt